CLINICAL TRIAL: NCT04932577
Title: Faecal Microbiota Transplantation to Prevent Complications, Progression and Mortality of Liver Cirrhosis
Brief Title: Faecal Microbiota Transplantation for Liver Cirrhosis
Acronym: CHiFT
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other); Aalborg University Hospital (Other); Odense University Hospital (Other); Hvidovre University Hospital (Other); Aalborg University (Other); Esbjerg Hospital - University Hospital of Southern Denmark (Other); Sjælland University Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1-10-72-302-20
Record Dates: First submitted 2021-05-26; First posted 2021-06-21 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2024-12

CONDITIONS: Liver Cirrhosis
Keywords: Hepatic encephalopathy; Ascites; Gastrointestinal bleeding; Spontaneous bacterial peritonitis; Hepatorenal syndrome; Alcoholic hepatitis
MeSH Terms: conditions — Liver Cirrhosis; Hepatic Encephalopathy; Ascites; Gastrointestinal Hemorrhage; Hepatorenal Syndrome; Hepatitis, Alcoholic | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Faecal microbiota transplantation (Experimental): The patients will receive three applications of FMT consisting of 50 g cryopreserved, homogenized faeces from healthy donors. The faecal material will be dispensed into double-coated, acid-resistant enterocapsules or cryobags. Faeces will be screened according to international guidelines.
  Interventions: Biological: Faecal microbiota transplantation
- Placebo (Placebo Comparator): The placebo products is produced from a suspension of glycerol, saline and food colouring and cannot be distinguished from the active FMT products.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Faecal microbiota transplantation — All participant will receive three applications of either FMT or placebo and afterwards followed for 1 year.
  Other Names: FMT
  Arms: Faecal microbiota transplantation
Biological: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose is to investigate the effect of faecal microbiota transplantation (FMT) on complications, progression, and mortality of patients with liver cirrhosis. Further, the investigators want to examine the impact of FMT on the gut microbiota, gut barrier function, systemic inflammation, and immune function.

DETAILED DESCRIPTION:
Patients with liver disease have a disturbed gut microbiota. This is often associated with disease progression and development of complications, so-called episodes of decompensation. In this trial, we will change the microbiota of these patients by transferring a healthy microbiota through faeces from a healthy donor, a procedure known as faecal microbiota transplantation (FMT). We will examine the effect of FMT on the prognosis and disease progression of the patients. Further, we will examine the mechanistic effects of FMT. We will at random divide 220 patients admitted with decompensation of liver cirrhosis evenly into two groups. One group will receive FMT and the other group will receive placebo. After the treatment, we will follow the patients for one year and examine disease progression as well as changes in their gut microbiota, gut barrier, and immune function.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years
* Liver cirrhosis with Child-Pugh ≤ 12
* Acute decompensation requiring intervention (ascites, gastrointestinal bleeding, infections leading to progressive liver failure, overthepatic encephalopathy, alcoholic hepatitis)

Exclusion Criteria:

* More than one organ failure defined by CLIF-SOFA score
* Untreated malignancy apart from non-melanoma skin cancer
* Untreated viral hepatitis
* HIV
* Inflammatory bowel disease
* Celiac disease
* Clostridioides Difficile infection
* Pregnancy
* Unable to participate based on medical judgement

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Time to death or new episode of acute decompensation requiring intervention in FMT versus placebo-treated patients. | 1 year
  Using data from the patient journals, we will be able to examine the exact time to event in each of the patients. To compare the two groups, hazard ratios will be calculated.

SECONDARY OUTCOMES:
Time to death or new episode of acute decompensation requiring intervention in FMT versus placebo-treated patients at 3 months and 6 months of follow-up. | 3 months, 6 months
  Using data from the patient journals, we will be able to examine the exact time to event in each of the patients. To compare the two groups, hazard ratios will be calculated.
Number of new decompensations and deaths during follow-up in the FMT versus the placebo-treated patients. | 1 year
  Incidence rates will be compared between the groups.
Time to death in FMT versus placebo-treated patients. -treated patients at 3 months and 6 months of follow-up. | 1 year, 6 months, 3 months
  Using data from the patient journals, we will be able to examine the exact time to event in each of the patients. To compare the two groups, hazard ratios will be calculated.
Change in gut microbiota beta-diversity (Bray-Curtis index) during one year in FMT versus placebo-treated patients by shotgun metagenomic sequencing. | 1 year, 6 months, 3 months
  In stool and saliva samples collected before and at 5 time points following the intervention, we will measure the gut microbiota composition.
Change in plasma concentration of gut translocation markers; lipopolysaccharide binding protein, soluble CD14, fatty acid binding protein 1 during one year in FMT versus placebo-treated patients by ELISA. | 1 year, 6 months, 3 months
  In blood samples collected at baseline and at follow-up visits, we will measure these plasma proteins by ELISA.
Change in plasma and stool concentration of pro- and antiinflammatory cytokines; IL-6, IL-1beta, TNF-alpha, IL-8, IL-10 in response to the intervention by luminex. | 1 year, 6 months, 3 months
  In blood and stool samples collected at baseline and at follow-up visits, we will measure these plasma proteins by luminex.
Change in disease severity in FMT- versus placebo-treated patients. | 3 months, 6 months, 1 year.
  The disease severity will be measured with Model for Endstage Liver Disease (MELD) (range 6-40). A high score reflects poor prognosis.
Change in disease severity in FMT- versus placebo-treated patients. | 3 months, 6 months, 1 year.
  The disease severity will be measured with Child-Pugh score (range 5-15). A high score reflects poor prognosis.
Change in disease severity in FMT- versus placebo-treated patients. | 3 months, 6 months, 1 year.
  The disease severity will be measured with CliF-C Acute decompensation scores (range 0-18). A high score reflects poor prognosis.
Change in metabolic liver function in FMT- versus placebo-treated patients. | 3 months, 6 months, 1 year.
  The metabolic liver function will be measured by the aminopyrine breath test
Change in liver stiffness in FMT- versus placebo-treated patients. | 3 months, 6 months, 1 year.
  Liver stiffness will be measured by liver elastography.
Change in the Liver Frailty Index in FMT- versus placebo-treated patients. | 3 months, 6 months, 1 year.
  The Liver Frailty index (grip strength, chair stands, and balance testing) will be calculated and the index will be compared between the treatment groups. A higher LFI indicates more frailty.
Change in body composition in FMT- versus placebo-treated patients. | 3 months, 6 months, 1 year.
  Body composition will be measured by bioimpedance.
Change in cognitive function as measured by continuous reaction time in FMT- versus placebo-treated patients. | 3 months, 6 months, 1 year.
  The cognitive function will be measured with continuous reaction time.
Change in cognitive function in FMT- versus placebo-treated patients. | 3 months, 6 months, 1 year.
  The cognitive function will be measured with the portosystemic encephalopathy syndrome test.
Change in quality adjusted life years (QALY´s) to evalute health care related costs in FMT- versus placebo-treated patients | 1 year
  By using the quality-of-life questionnaire (EQ-5D-5L) a single index will be calculated and used to calculate QALY's.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Hepatology and Gastroenterology, Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stoy S, Eriksen LL, Lauszus JS, Damsholt S, Baunwall SMD, Erikstrup C, Vilstrup H, Jepsen P, Hvas C, Thomsen KL. Cirrhosis and Faecal microbiota Transplantation (ChiFT) protocol: a Danish multicentre, randomised, placebo-controlled trial in patients with decompensated liver cirrhosis. BMJ Open. 2025 Feb 12;15(2):e091078. doi: 10.1136/bmjopen-2024-091078. PMID 39938959